CLINICAL TRIAL: NCT01502202
Title: A Randomized Placebo-controlled Phase II Study of Intercalated Administration of Pemetrexed/Cisplatin With Iressa® (Gefitinib) or Placebo as First-line Treatment of Stage IIIB/IV Lung Adenocarcinoma in Never-smokers
Brief Title: Intercalated Administration of PamCis With Gefitinib or Placebo as First Line Lung Adenocarcinoma in Never Smokers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Jin Soo Lee, Principal Investigator, National Cancer Center, Korea
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCCCTS-11-581
Record Dates: First submitted 2011-12-22; First posted 2011-12-30 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Non Small Cell Lung Cancer; Adenocarcinoma
Keywords: lung adenocarcinoma; never smoker; 1st line treatment; Intercalation administration; Gefitinib; never smokers
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma; Adenocarcinoma of Lung | interventions — Gefitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study arm (Active Comparator): Pemetrexed plus Cisplatin plus Gefitinib
  Interventions: Drug: Gefitinib; Drug: Pemetrexed plusCIsplatin
- Placebo arm (Placebo Comparator): Pemetrexed plus Cisplatin plus Placebo
  Interventions: Drug: Placebo; Drug: Pemetrexed plusCIsplatin

INTERVENTIONS:
Drug: Gefitinib — Gefitinib 250mg, per PO. daily, D 5-18 (during 14 days)
  Other Names: AP-G
  Arms: Study arm
Drug: Placebo — Placebo 1 tablet, per PO, Daily on D 5-18 (during 14 days)
  Other Names: AP-P
  Arms: Placebo arm
Drug: Pemetrexed plusCIsplatin — Pemetrexed 500mg/m2 on D1 plus Cisplatin 75mg/m2 on D1 every 3 weeks maximum 9 cycles
  Other Names: Standard chemotherapy

SUMMARY:
Intercalated administration of Iressa® (gefitinib) on days 5-18 of chemotherapy cycle improve the efficacy of Pemetrexed/platinum regimen given as first-line treatment for never-smokers with advanced (stage IIIB/IV) lung adenocarcinoma.

DETAILED DESCRIPTION:
Investigators believe this PFS curve crossing-over in both IPASS and First-SIGNAL study is mainly due to early progression of EGFR mutation-negative tumors after gefitinib alone. Taken together with the FASTACT trial results, this PFS curve crossing-over may well be averted if effective chemotherapy is given together with gefitinib in a most optimum timing and sequence. Apparently, timing of EGFR-TKI administration within chemotherapy cycles is very critical, as shown in OSI 9774 trial.

In this placebo-controlled randomized phase II, Investigators propose to give gefitinib on days 5-18 of a 3-weekly chemotherapy cycle of pemetrexed/cisplatin to avoid any potential overlap of EGFR-TKI effects on chemotherapy or vice versa. Investigators would like to generate promising pilot data, which warrants a large phase III trial. Investigators hope to show that intercalated administration of Iressa® (gefitinib) and Pemetrexed/platinum regimen improves the outcome of never-smokers with advanced (stage IIIB/IV) lung adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of adenocarcinoma of lung with or without BAC features; however, adenocarcinoma combined with other histology, such as small cell carcinoma or squamous carcinoma, is not allowed.
2. Stage IIIB (not amenable for radical loco-regional therapy) or stage IV (metastatic) patients according to the 7th TNM staging system
3. Age 18-75
4. Never-smoking defined as not more than 100 cigarettes during the lifetime
5. ECOG performance status of 0-2
6. Good organ function
7. The presence of CNS metastases is not considered as an exclusion criterion, provided that there is good control of the symptoms with corticosteroids
8. Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policy of the hospital. The only approved consent form is attached to this protocol

Exclusion Criteria:

1. Patients with prior exposure to agents directed at the HER
2. Patients with prior chemotherapy or therapy with systemic anti-tumour therapy for advanced disease.
3. Lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome, or inability to take oral medication, or have active peptic ulcer disease.
4. Known severe hypersensitivity to gefitinib or to any of the study drugs.
5. Any evidence of clinically active interstitial lung disease
6. Concomitant use of phenytoin, carbamazepine, rifampicin, barbiturates, or St John's Wort
7. Prior invasive malignancies 3 years prior to study entry except adequately treated cutaneous basal cell carcinoma or uterine cervix in situ cancer
8. As judged by the investigator, any evidence of severe or uncontrolled systemic disease
9. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the study
10. Treatment with a non-approved or investigational drug within 30 days before Day 1 of study treatment.
11. Pregnancy or breast-feeding (women of child-bearing potential).
12. Sexually active males and females (of childbearing potential) unwilling to practice acceptable methods of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-08 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
To compare progression-free survival | minimum 1-year follow-up
  from date of randomization until the date of first documented progression or death from any case.
  Assessed minimum 1 years.

SECONDARY OUTCOMES:
To compare objective response rate (CR+PR) | minimum 1-year follow-up
  every 9 weeks until PD
To compare duration of response. | minimum 1-year follow-up
To compare non progression rate (CR+PR+SD) at 16 weeks. | at 16 weeks
To compare overall survival. | minimum 1-year follow-up
To compare number of Grade 3/4 Adverse Events | average up to 1 year
  Participants will be followed for the duration of chemotherapy. CTCAE version 4.0
To assess biomarker | minimum 1-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jin Soo Lee, M.D. PhD., Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang-si, Gyenggido, South Korea